CLINICAL TRIAL: NCT02022254
Title: An Open-label, One-sequence Cross Over, Single Centre Trial, Investigating the Influence of Semaglutide on Pharmacokinetics and Pharmacodynamics of Warfarin and Pharmacokinetics of Metformin in Healthy Subjects
Brief Title: Influence of Semaglutide on Pharmacokinetics and Pharmacodynamics of Warfarin and Pharmacokinetics of Metformin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-3817; 2012-005072-33 (EudraCT Number); U1111-1136-6442 (Other: WHO)
Record Dates: First submitted 2013-12-16; First posted 2013-12-27 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Metformin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semaglutide administrations (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo; Drug: metformin; Drug: warfarin

INTERVENTIONS:
Drug: semaglutide — Subjects will initiate treatment with 0.25 mg for the first four weeks followed by dose doubling every four weeks up to a dose of 1.0 mg.
Drug: placebo — Semaglutide placebo will be administered s.c.
Drug: metformin — For oral administration twice daily, in two periods, each of 3.5 days duration. The first period is initiated before semaglutide treatment and the second period is initiated at the end of semaglutide treatment.
Drug: warfarin — For oral administration, given as a single dose. The first dose is given before semaglutide treatment and the second dose is given at the end of semaglutide treatment.

SUMMARY:
This trial is conducted in Europe and Asia. The aim of the trial is to investigate the influence of semaglutide on pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of warfarin and pharmacokinetics of metformin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age between 18 and 55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 23 and 30 kg/m^2 (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearingpotential and not using adequate contraceptive methods for the duration of the trial and for 5 weeks following the last dose of semaglutide. Adequate contraceptive measures are implants, injectables, combined oral contraceptives, hormonal intrauterine device, sexual abstinence or vasectomised partner
* Any clinically significant disease history, in the opinion of the investigator, or systemic or organ disease including: pulmonary, gastrointestinal, hepatic, neurologic, renal, genitourinary and endocrine, dermatologic or hematologic diseases
* Use of prescription or non-prescription systemic or topical medicinal products (including routine or non-routine vitamins or herbal products, but excluding paracetamol and contraceptives) within 3 weeks (or within 5 half-lives of the medicinal product, whichever is longest) prior to Visit 2
* Smoking, drug or alcohol abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12-17 (Actual); Primary Completion 2014-08-28 (Actual); Study Completion 2014-08-28 (Actual)

PRIMARY OUTCOMES:
Area under the metformin plasma concentration-time curve | During a dosing interval (0-12 hours) after the last of 7 repeated doses of metformin without semaglutide exposure (Day 4) and at semaglutide steady state (Day 104)
Area under the S-warfarin plasma concentration-time curve | From time 0 to 168 hours after a single dose of warfarin without semaglutide exposure (Day 11) and at semaglutide steady state (Day 111)
Area under the R-warfarin plasma concentration-time curve | From time 0 to 168 hours after a single dose of warfarin without semaglutide exposure (Day 11) and at semaglutide steady state (Day 111)

SECONDARY OUTCOMES:
Maximum observed metformin plasma concentration at steady state | From dosing until 30 hours after the last of 7 repeated doses without semaglutide exposure and at semaglutide steady state (metformin administration on Days 4 and 104)
Maximum observed S-warfarin plasma concentration after single dose | (0-168 hours) after a single dose of warfarin without semaglutide exposure and at semaglutide steady state (warfarin administrations on Days 11 and 111)
Maximum observed R-warfarin plasma concentration after single dose | (0-168 hours) after a single dose of warfarin without semaglutide exposure and at semaglutide steady state (warfarin administrations on Days 11 and 110)
Incremental area under the INR (international normalised ratio) -curve | From 0 to 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Result] Hausner H, Derving Karsbol J, Holst AG, Jacobsen JB, Wagner FD, Golor G, Anderson TW. Effect of Semaglutide on the Pharmacokinetics of Metformin, Warfarin, Atorvastatin and Digoxin in Healthy Subjects. Clin Pharmacokinet. 2017 Nov;56(11):1391-1401. doi: 10.1007/s40262-017-0532-6. PMID 28349387
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com